CLINICAL TRIAL: NCT07400822
Title: İnme Sonrası Yutma Bozukluğu Gelişen Hastalara Erken Dönemde Verilen Ekşi Sıvının Yutma Fonksiyonu Üzerine Etkisinin Değerlendirilmesi
Brief Title: Effect of Sour Taste on Swallowing Function of Patients With Dysphagia After Acute Ischemic Stroke: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AYFER GUNES (Other)
Collaborators: Trakya University (Other)
Responsible Party: Sponsor-Investigator, AYFER GUNES, Dr. (PhD), Register Nurse, Trakya University
Organization: Trakya University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021/214
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Cerebrovascular Accident; Dsyphagia After Stroke
Keywords: Stroke, dysphagia, sour liquid, swallowing function, nurse
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Other): The participants were informed about the research process during the first meeting. Control group patients were administered 4 ml of room temperature water during the initial consultation, under the supervision of a physician, before breakfast, lunch, and dinner. According to the GUSS screening test, patients with severe dysphagia were given 4 ml of water drop by drop with a syringe, in a manner tolerable to the patient, together with the physician, over approximately 15-20 minutes. Stroke patients with severe dysphagia, unable to swallow, had the 4 ml of water administered drop by drop but it flowed out of their mouths as saliva. This procedure was continued for seven days .Patients with dysphagia who had acute ischemic stroke in the control group was evaluated at the first day visit, on the day 7, and day 30. The initial visit and day 7 evaluations were conducted in a clinical setting because the patients were receiving treatment at the neurology clinic.
  Interventions: Other: Control
- Sour Taste (Experimental): The participants were informed about the research process during the first meeting. Intervention group patients were administered 4 ml of freshly squeezed lemon juice with a hydrogen power (pH) of 2.8 at room temperature under medical supervision before breakfast, lunch, and dinner. According to the GUSS screening test, patients with severe dysphagia were given 4 ml of lemon juice drop by drop with a syringe, in a manner tolerable to the patient, together with the physician, over approximately 15-20 minutes. Patients with severe dysphagia, due to their inability to swallow, had the 4 ml of lemon juice administered drop by drop, but it flowed out of their mouths as saliva. This application continued for seven days.Patients with dysphagia who had acute ischemic stroke in the control group was evaluated at the first day visit, on the day 7, and day 30. The initial visit and day 7 evaluations were conducted in a clinical setting because the patients were receiving treatment at the neurolo
  Interventions: Other: sour taste

INTERVENTIONS:
Other: sour taste — Sour taste stimulation using freshly squeezed lemon juice administered orally.
  Arms: Sour Taste
Other: Control — Room-Temperature Water Administration
  Arms: control

SUMMARY:
This randomized controlled study was designed to determine the Effect of Sour Taste on Swallowing Function of Patients with Dysphagia After Acute Ischemic Stroke The study was conducted between july 2021 and november 2022 with 95 patients diagnosed with Acute Ischemic Stroke (47 intervention, 48 control) at the neurology clinic and outpatient clinic of a university hospital in Edirne. Data were collected using the Personal Information Form, the Gugging Swallowing Screening Test (GUSS), and the National Institutes of Health Stroke Scale (NIHSS).

DETAILED DESCRIPTION:
This study was designed to evaluate the effect of sour taste on swallowing function of patients who developed dysphagia after ischemic stroke.The study sample consisted of patients (n=95) diagnosed with ischemic stroke and had impaired swallowing function hospitalized in a neurology clinic of a university hospital. Patients in the intervention group were given 4 ml of lemon juice (pH=2.8) at room temperature before breakfast, lunch, and dinner, while patients in the control group were given 4 ml of water at room temperature at the same time periods. Patients' swallowing function and stroke severity were assessed on the 7th and 30th days. Data were collected using the Personal Information Form, the Gugging Swallowing Screening Test (GUSS), and the National Institutes of Health Stroke Scale (NIHSS).

Financial Support:The present study was supported by the Research Fund of Trakya University. Project No:2021/214

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with a confirmed diagnosis of ischemic stroke
* Within the first 72 hours after diagnosis
* Developed dysphagia
* Who could understand and cooperate
* Patients who volunteer signed an informed consent

Exclusion Criteria:

* Patients with cerebral hemorrhage or other neurologic disorders
* Patients with severe stroke and high NIHSS scores
* Who were likely to experience severe dysphagia
* Patients who do not volunteer to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
GUSS Swallowing scores and NIHSS Scores | one month
  Change in the mean scores of the GUSS swallowing scores and NIHSS Scores of the patients at the first interview, on the 7th day and on the 30th day.

CONTACTS AND LOCATIONS:
Overall Officials: Ayfer Gunes, PhD, RN., Principal Investigator — Trakya University Medical Research and Application Centre, Department of Neurology
Locations (1):
- Trakya University Medical Research and Application Centre, Edirne, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided